CLINICAL TRIAL: NCT04564365
Title: Influence of Beta-Blockers on Prognosis in Patients With Acute Myocardial Infarction Complicated With Normal Ejection Fraction
Brief Title: The Contemporary Role of Beta Blockers in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Professor, Chongqing Medical University
Other Study IDs: 2020-09-22
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-06

CONDITIONS: Acute Coronary Syndrome
Keywords: left ventricular ejection fraction; acute myocardial infarction; beta-blocker
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with beta-blocker
  Interventions: Drug: beta-blocker
- without beta-blocker

INTERVENTIONS:
Drug: beta-blocker — To investigate the relationship between the use of beta blockers and prognosis in patients with normal ejection fraction after acute myocardial infarction
  Groups: with beta-blocker

SUMMARY:
The use of beta blockers after acute myocardial infarction is a core component of drug therapy, but evidence is primarily derived from patients who did not receive reperfusion therapy and secondary prophylaxis.In contemporary times, the prognostic value of beta blockers in patients with acute myocardial infarction has been questioned, particularly in patients without reduced heart failure/ejection fraction after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of acute myocardial infarction was clear and the left ventricular ejection fraction was normal

Exclusion Criteria:

* History of heart failure Died in hospital

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient had normal left ventricular ejection fraction (LVEF≥50%) after acute myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-11-25 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
mortality | the median time of 8 months
  all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated Hospital of Chongqing Medical University, Chongqing, China